CLINICAL TRIAL: NCT05354440
Title: Long-Term Prospective Post Marketing Clinical Follow Up for Evaluation of the BioProtect Balloon Implant System
Brief Title: Post Marketing Clinical Follow Up of the BioProtect Balloon Implant System
Acronym: CLP-10441
Status: Active, not recruiting | Type: Observational
Sponsor: BioProtect (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-10441
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Long-Term Prospective Post Marketing Clinical Follow Up for Evaluation of the BioProtect Balloon Implant™ System

DETAILED DESCRIPTION:
Multi-center, long-term, prospective, observational study for assessment of late rectal toxicity and quality of life in prostate cancer subjects undergoing radiotherapy by means of IMRT following implantation of the BioProtect Balloon Implant System.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has previously participated in the BP-007 clinical study and completed their IMRT treatment.
2. Subject agrees to complete all required follow-up visits.
3. Subject provides written Informed Consent prior to any study related procedure

Exclusion Criteria:

1. Subject who completed 48 months of follow-up in the BP-007 study.
2. Subjects who are receiving at the time of the study, any other investigational agents/ devices.
3. Subjects unwilling and/or unable to comply with the provisions of the study protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate Cancer
Study Population: Subjects who previously participated in the BP-007 clinical study
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Long Term Rectal And Urinary Toxicity and Quality of Life | 48 months
  Long-term safety as assessed by incidence of urinary and bowel toxicities.

CONTACTS AND LOCATIONS:
Locations (6):
- St Luke's Radiation Oncology, Dublin, Ireland
- Israel (2):
  - Assuta Ashdod medical center, Ashdod
  - Rabin Medical Center, Petah Tikva
- Maastricht radiation oncology, Maastricht, Netherlands
- Institute of Maria Skłodowska - Curie, Warsaw, Poland
- Cuf Porto institution, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No